CLINICAL TRIAL: NCT06040177
Title: Efficacy and Safety of SBRT Combined With Cardonilizumab and Lenvastinib in the Treatment of Unresectable Hepatocellular Carcinoma With Portal Vein Tumor Thrombus#a Prospective, Multicenter, Single-arm Clinical Study
Brief Title: Efficacy and Safety of SBRT Combined With Cardonilizumab and Lenvastinib in the Treatment of Unresectable Hepatocellular Carcinoma With Portal Vein Tumor Thrombus
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jie Ma, Clinical Professor, First Affiliated Hospital of Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GuangxiMUMJ1
Record Dates: First submitted 2023-07-13; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Hepatocellular Carcinoma Non-resectable; Portal Vein Tumor Thrombus; Immune Checkpoint Inhibitors
Keywords: Hepatocellular Carcinoma; portal vein tumor thrombus; Immune Checkpoint Inhibitors; Efficacy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT+cardonilizumab+lenvastinib Group (Experimental): Renvatinib: 8mg (weight <60kg) or 12mg (weight ≥60kg) once a day until disease progression, intolerable toxicity Radiation therapy: Stereotactic radiotherapy (5-8Gy*5F) for portal vein thrombus within 21 days after entry Cadonilimab will be administered within 2 weeks after the completion of the radiotherapy treatment once every 3 weeks (Q3W), for up to 2 years
  Interventions: Drug: Cadonilimab; Radiation: Stereotactic radiotherapy; Drug: Renvatinib

INTERVENTIONS:
Drug: Cadonilimab — Cadonilimab will be administered within 2 weeks after the completion of the radiotherapy treatment once every 3 weeks (Q3W), for up to 2 years
  Other Names: AK104
Radiation: Stereotactic radiotherapy — Radiation therapy: Stereotactic radiotherapy (5-8Gy*5F) for portal vein thrombus within 21 days after entry
Drug: Renvatinib — Renvatinib: 8mg (weight <60kg) or 12mg (weight 60kg) once a day until disease progression, intolerable toxicity

SUMMARY:
This study is a single-arm, multicenter clinical study to evaluate the efficacy and safety of SBRT combined with cardonilizumab and lenvastinib in the treatment of unresectable hepatocellular carcinoma with portal vein tumor thrombus

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years old;
2. Eastern Cooperative Oncology Group (ECOG) -Performance Status(PS):0-2 points；
3. Hepatocellular carcinoma was diagnosed according to histopathology or the 2022 diagnostic criteria for primary liver cancer；
4. Expected survival period≥3 months;
5. Liver function grade Child-Pugh A or better grade B (7 points);
6. At least one measurable lesion:

   Liver lesion ① The Lesion can be accurately measured at least in the range of 1.0cm;

   ② The Lesion is suitable for repeated measurement;
   * The lesion shows enhanced intratumoral arteries on computed tomography (CT) or magnetic resonance imaging (MRI); Non-liver lesion In at least one dimension, the short axis of lymphadenopathy (LN) is≥1.5cm. Longest diameter of non-nodular lesions is≥1.0cm
7. The Barcelona liver cancer staging system is stage C (BCLC-C), which meets one of the following conditions:

(1) Liver tumor can be resected, which is combined with Vp 3-4 portal vein cancer thrombus; (2) Liver tumor is unresectable or has distant metastasis, and is combined with Vp1-4 type portal vein cancer thrombus; 8. The patient had not received prior systemic therapy including sorafenib, lenvatinib, chemotherapy; 9. The patient had previously received locoregional therapy (including radiofrequency or ablation therapy, percutaneous ethanol or acetic acid injection, cryotherapy, high intensity focused ultrasound, hepatic artery chemoembolization, hepatic artery embolization, etc., and the local treatment area had definite progression (according to RECIST v1.1 criteria); 10. Baseline blood routine and biochemical indicators meet the following criteria: Hemoglobin≥90g / L; Absolute neutrophil count (ANC)≥1.5× 10 ^ 9 / L; Platelet≥75×10 ^ 9 / L; ALT,AST ≤3×upper normal value (ULN); Serum total bilirubin ≤ 1.5 ×ULN; Serum creatinine ≤1.5 × ULN; Serum albumin was used for≥30g / L.

Exclusion Criteria:

1. Patients diagnosed with hepatobiliary duct cell carcinoma, mixed cell carcinoma, or fibrolaminar cell carcinoma；
2. Patients with a history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation or planned transplantation；
3. Patients have hepatic encephalopathy (West Haven Standard Grade III, Level IV) or have moderate or severe ascites (i.e., patients requiring therapeutic puncture drainage) or have uncontrolled pleural or pericardial effusion；
4. Patients have symptomatic, untreated, or progressive central nervous system (CNS) or leptomeningeal metastases.If all the following criteria are met, asymptomatic subjects with treated CNS lesions can be enrolled.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | Up to approximately 2 years
  ORR is proportion of patients with complete response(CR) or partial response(PR) assessed by investigators according to RECIST v1.1.

SECONDARY OUTCOMES:
3-month PFS rate | Up to approximately 2 years
  3-month PFS rate is the percentage of patients whose disease has not progressed within 3 months.
progression-free survival (PFS) | Up to approximately 2 years
  Progression-free survival (PFS) is defined as the time from the first dose of Cadonilimab until documentation of PD (as per RECIST v1.1) or death due to any cause, whichever occurs first.
Disease control rate (DCR) | Up to approximately 2 years
  DCR is proportion of patients with complete response, partial response or stable disease assessed by investigators according to RECIST v1.1.
Duration of response (DOR) | Up to approximately 2 years
  Duration of Response (DOR) is defined as the time between the first assessment of a tumor as Complete Response（CR）or Partial Response（PR）and the first assessment of Progressive Disease (PD) or death from any cause.
Overall Survival (OS) | Up to approximately 2 years
  Overall survival (OS) is defined as the time from the first dose of Cadonilimab until death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China

REFERENCES:
- [Derived] Mo N, Hu K, Zeng Z, Yang L, Fang Y, Zeng J, Li Y, Yang Z, Tang J, Zhang T, Ma F, Liu C, Zheng H, Qiu J, Jiang Y, Lv Y, Liang L, Huang X, Liao X, Wang Y, Lu X, Ning L, Lao Guo S, Ma J, Wang R. Stereotactic body radiation therapy combined with cadonilimab and lenvatinib in the treatment of hepatocellular carcinoma with Vp3 or Vp4 portal vein tumor thrombus: a prospective, multicenter, single-arm, phase II clinical trial. Front Immunol. 2025 Nov 10;16:1687344. doi: 10.3389/fimmu.2025.1687344. eCollection 2025. PMID 41293180